CLINICAL TRIAL: NCT02452593
Title: Randomized Trial of Tibial Nerve Stimulation Versus Pelvic Floor Exercises for Treatment of Overactive Bladder, Urge and Mixed Urinary Incontinence
Brief Title: Randomized Trial of Tibial Nerve Stimulation Versus Pelvic Floor Exercises for Treatment of Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Magda da Silva Aranchipe, Researcher, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UFRGSDGO
Record Dates: First submitted 2015-04-08; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Urge Incontinence
Keywords: incontinence; pelvic floor exercises; neuromodulation
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Tibial Nerve Stimulation" (Active Comparator): This group will do transcutaneous electrical stimulation of the tibial nerve at home.
  Development of an innovative portable equipment, with domestic technology for home application of the posterior tibial nerve stimulation technique using the type SSP surface electrodes (Silver Spike Point). Frequency: 20 Hz, Pulse width: 200 us; duration: 15min daily
  Interventions: Other: "Tibial stimulation" and "pelvic floor exercises"
- "Pelvic Floor Exercises" (Active Comparator): This group will make pelvic muscle training 3 times a day . In decubit dorsal posture, legs flexed and abductee. Perform pelvic floor contractions keeping 2 seconds and relaxing 4 seconds for 10 times, and contractions keeping 4 seconds and relaxing 8 seconds for 10 times.
  Interventions: Other: "Tibial stimulation" and "pelvic floor exercises"

INTERVENTIONS:
Other: "Tibial stimulation" and "pelvic floor exercises" — A group will make tibial nerve stimulation and the other will make pelvic floor training. After 8 weeks the patients exchanges their therapeutic approaches for over 8 weeks

SUMMARY:
Urinary incontinence is defined according to the International Continence Society as any involuntary loss of urine, which may bring several negative consequences on women's lives, and among incontinent women, about 50% have urinary incontinence, 30% mixed and 20% emergency.

The overactive bladder present in urge incontinence and mixed cause significant impacts on people's lives and has a prevalence of 16.5% in the US population.

Behavioral therapies, exercises the pelvic muscles and drugs are the main forms of treatment. Drug therapy using drugs which are not specific for the bladder and are associated with many unwanted systemic side effects.

The results obtained by researchers in several countries using conservative techniques in the treatment of patients with urinary incontinence are encouraging and this study aims to evaluate carefully and systematically the effectiveness of tibial stimulation technique.

Importantly, also, that conservative techniques have lower cost than the surgical treatment and have virtually no side effects as most of the drugs used in the pharmacological treatment of female urinary incontinence.

DETAILED DESCRIPTION:
Goal

Development of instrumentation for home treatment of overactive bladder and urgency / mixed incontinence using tibial stimulation and pelvic floor exercises.

Secondary objectives

* Development of an innovative portable equipment, with domestic technology for home application of the posterior tibial nerve stimulation technique using the type SSP surface electrodes (Silver Spike Point).
* Comparison of the effectiveness of tibial stimulation techniques and pelvic floor exercises in the treatment of overactive bladder and urgency / mixed incontinence.

Design Randomized Clinical Trial

Sample Women over the age of 18, complaining of urinary incontinence Urgency or Mixed (with main urgency component), catered in Urogynecology Ambulatory of Hospital de Clinicas de Porto Alegre.

ELIGIBILITY:
Inclusion Criteria:

- Women with Urinary Incontinence of Urgency or Mixed older than 18 years

Exclusion Criteria:

* Presence Of vaginal or urinary infection
* Not understand or sign the informed consent
* Not understand or are unable to perform the proposed treatment
* Pregnancy or the postpartum period covering the period up to 6 months after delivery
* Women in previous use of chronically used drugs (antidepressants, diuretics, and others) that can evidently alter the urinary function.
* Stress Urinary Incontinence of pure or mixed incontinence with a predominance of Stress component neurogenic bladder
* Use of Botox® in the bladder or pelvic muscles in the last year
* Use Interstim® or Bion®
* Use pacemaker or implantable defibrillator
* Current use of TENS in the pelvic region, lower back or legs
* Previous use of percutaneous tibial stimulation
* Drug / experimental devices in the past 4 weeks,
* Participation in any clinical research involving or affecting the urinary or renal function in the last 4 weeks.
* Pelvic radiotherapy;
* Changes in sensibility Lower Limb;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Urinary incontinence | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Geraldo Dr Ramos, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil